CLINICAL TRIAL: NCT02625376
Title: Influence of Resveratrol and Resvega Versus Placebo on Incidence of Bilateralisation of Exudative AMD: a Double Masked Prospective Study.
Brief Title: Resveratrol for Exudative Age-Related Macular Degeneration
Acronym: AGED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AGED/EudraCT : 2015-001577-41
Record Dates: First submitted 2015-08-06; First posted 2015-12-09 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: AMD; Age-related Macular Degeneration; Choroidal Neovascularisation
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trans-Resveratrol (Experimental): capsule of 250 mg of resveratrol. two capsules daily : one in the morning and evening for 24 months
  Interventions: Dietary Supplement: Trans-Resveratrol
- Resvega (Active Comparator): capsule composed of antioxydant, omega 3, carotenoid, 15 mg of resveratrol, zinc and copper.
  two capsules daily : one in the morning and evening for 24 months
  Interventions: Dietary Supplement: Resvega
- Placebo (Placebo Comparator): capsule of medium chain triglyceride. two capsules daily : one in the morning and evening for 24 months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Resvega — Dietary supplementation with Resvega BD
  Arms: Resvega
Dietary Supplement: Trans-Resveratrol — Dietary supplementation with resveratrol 250 mg BD
  Arms: Trans-Resveratrol
Dietary Supplement: placebo — Dietary supplementation with a placebo BD
  Arms: Placebo

SUMMARY:
This is an interventional, prospective, randomized, comparative monocentric study aiming to evaluate the safety and efficacy of Resveratrol to reduce the progression of exudative Age-Related Macular Degeneration.

DETAILED DESCRIPTION:
Interventional, prospective, randomized, comparative monocentric study aiming to evaluate the safety and efficacy of Resveratrol to reduce the progression of exudative Age-Related Macular Degeneration.

Comparison of incidence of choroidal neaovascularization between each study group will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 55 or more with unilateral exudative AMD
* Visual acuity less or equal to 20/25 in the most affected eye

Exclusion Criteria:

* Allergy to an investigational product
* atrophic Age-Related Macular Degeneration or age related maculopathy
* significant media opacities
* Other retinal pathology (diabetic retinopathy, high myopia, retinal dystrophy)
* Recent Cataract surgery
* Previous history of vitrectomy
* Acute or chronic severe organ failure
* Present participation in other clinical research study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Comparaison of incidence of choroidal neovascularization between resveratrol group and placebo group at 24 months | 24 months
  What is the influence of the daily intake of 500 mg of resveratrol on the incidence of neovascularization of the second eye?

SECONDARY OUTCOMES:
Comparaison of incidence of choroidal neovascularization between Resvega group and placebo group at 24 months | 24 months
  What is the influence of the daily intake resvega on the incidence of neovascularization of the second eye?

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEVEZIEL, MD, PhD, Principal Investigator — Dpt of Ophthalmology, University Hospital of Poitiers, France
Locations (1):
- CHU de Poitiers - Ophtalmology, Poitiers, France

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300